CLINICAL TRIAL: NCT05786079
Title: Effects of Footstrike Transition on Tibial Stress Fracture Risk Using Musculoskeletal Simulation, Finite Element Analysis and Probabilistic Modelling - a Pilot Study
Brief Title: Effects of Footstrike Transition on Tibial Stress Fracture Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Principal Investigator and Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Footstrike tibial stress
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Tibial Stress Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Footstrike modification (Experimental)
  Interventions: Behavioral: Footstrike modification
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Footstrike modification
  Arms: Footstrike modification
Behavioral: Control
  Arms: Control

SUMMARY:
Biomechanical literature suggests that runners who utilize a mid or forefoot strike pattern may suffer from a reduced incidence of chronic injuries compared to a rearfoot strike. This investigation examined the effects of a 10-week footstrike transition intervention on tibial stress fracture risk in runners.

ELIGIBILITY:
Inclusion Criteria:

* Recreational runner
* 3-years minimum of running experience
* Injury free for 12-months

Exclusion Criteria:

* Injury at baseline

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Stress fracture probability | Baseline
  Probability of stress fracture quantified using a probabilistic modelling approach.
Stress fracture probability | 10-weeks
  Probability of stress fracture quantified using a probabilistic modelling approach.

SECONDARY OUTCOMES:
Three-dimensional tibial loading | Baseline
  Forces applied to the tibia, measured using musculoskeletal simulation.
Three-dimensional tibial loading | 10-weeks
  Forces applied to the tibia, measured using musculoskeletal simulation.
Tibial strain | Baseline
  Strains experienced by the tibial quantified using finite elements analysis.
Tibial strain | 10-weeks
  Strains experienced by the tibial quantified using finite elements analysis.

IPD SHARING:
Plan to Share IPD: No